CLINICAL TRIAL: NCT01308541
Title: A Randomized, Open-label, 3 Period Crossover Study to Characterize the Pharmacokinetics and Pharmacodynamics of LUSEDRA (Fospropofol Disodium) Injection Administered Either by Continuous Infusion or Bolus Compared With Continuous Infusion of Propofol Injectable Emulsion
Brief Title: A Study to Characterize Pharmacokinetics (PK) and Pharmacodynamics (PD) of LUSEDRA® Administered as Continuous Infusion or Bolus Compared With Continuous Infusion of Propofol Injectable Emulsion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E2083-A001-006
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Monitored Anesthesia Care
MeSH Terms: interventions — fospropofol; Propofol

ARMS (3):
- LUSEDRA (arm 1) (Active Comparator)
  Interventions: Drug: arm 1
- LUSEDRA (arm 2) (Active Comparator)
  Interventions: Drug: LUSEDRA
- Propofol (arm 3) (Active Comparator)
  Interventions: Drug: Propofol (arm 3)

INTERVENTIONS:
Drug: arm 1 — Bolus Dose: two bolus doses of 15.0 mg/kg (first dose) and 8.0 mg/kg (second dose), 40 minutes apart.
  Continuous Infusion Dose: Total dose of 42.0 mg/kg administered over 3 hours at an infusion rate of 0.40 mg/kg/min for 1 hour, followed by 0.20 mg/kg/min for 1 hour, followed by 0.10 mg/kg/min for 1 hour.
  Arms: LUSEDRA (arm 1)
Drug: LUSEDRA — Mode of administration: intravenous (IV).Continuous Infusion Dose: Total dose of 42.0 mg/kg administered over 3 hours at an infusion rate of 0.40 mg/kg/min for 1 hour, followed by 0.20 mg/kg/min for 1 hour, followed by 0.10 mg/kg/min for 1 hour.
  Arms: LUSEDRA (arm 2)
Drug: Propofol (arm 3) — Mode of administration: intravenous (IV). A loading dose administered at a constant infusion rate of 0.20 mg/kg/min (0.50 mL/kg/min) for 10 minutes, followed by a constant-rate 2-hour infusion at 0.10 mg/kg/min; total dose infused over 130 minutes is 14.0 mg/kg.
  Arms: Propofol (arm 3)

SUMMARY:
The purpose of this study is to explore the pharmacokinetics (PK) and pharmacodynamics (PD) of LUSEDRA® administered as a continuous infusion or bolus compared with continuous infusion of propofol injectable emulsion.

DETAILED DESCRIPTION:
The study is designed to explore the pharmacokinetics (PK) and the pharmacokinetic/ pharmacodynamic (PK/PD) relationship between PK-Bispectral Index (BIS) and PK-Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores following administration of LUSEDRA, administered as a bolus or by continuous infusion, with that of propofol injectable emulsion administered by continuous infusion, using compartmental modeling. The clinical practice of sedation spans an entire continuum of sedation, only a portion of which is currently addressed by the currently approved dose which is intended to provide a moderate level of sedation. Another goal of the current study is to support potential follow-up indications for fospropofol disodium, such as prolonged sedation in the Intensive Care Unit (ICU) and induction and maintenance of general anesthesia, which require higher doses. If successful, the data from this study would allow a direct comparison of propofol doses, delivered as fospropofol disodium or as propofol injectable emulsion, that provide the same sedation effect and directly compare concentration-effect relations of propofol liberated from fospropofol disodium with that delivered as propofol. The doses and infusion times for fospropofol disodium and propofol in this study were selected based on simulation results using an established PK/PD model developed from historical data. Data collected in the current study will be used to further refine the existing PK/PD model. To enhance the robustness of that model, the study design includes changes in dose over the duration of sedation in the three treatment groups.

ELIGIBILITY:
Inclusion:

* Nonsmoking male and female subjects, age >/= 18 to </= 45 years old at Screening.

Exclusion:

* Body mass index (BMI) >/= 30
* Subjects who smoke or have used nicotine or nicotine-containing products within 18 months of Screening and throughout the study
* Subjects with a known history of clinically significant drug or food allergies, including allergies to any ingredients in either medication (fospropofol disodium or propofol injectable emulsion) or presently experiencing significant seasonal allergy
* Subjects who are allergic to eggs, egg products, soybeans, or soy products
* Subjects having a past or current medical history of any respiratory illness including asthma or sleep apnea
* Subjects with disorders of fat metabolism, or who are predisposed to fat embolism, or who have other conditions in which lipid emulsions must be used carefully
* Subjects currently taking any medications including over-the-counter (OTC) medication (within 14 days prior to Baseline Period 1) with the exceptions of hormonal contraceptives and hormone replacement therapy, as long as the subject was on a stable dose of the same product for at least 12 weeks prior to dosing.
* Use of 1.0% lidocaine <1.0 mL for placement of all arterial lines is allowed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Arterial plasma levels of fospropofol and propofol during each treatment: | up to 480 minutes postdose

SECONDARY OUTCOMES:
PD effect during each treatment measured by continuous BIS recordings | up to 480 minutes postdose
PD effect during each treatment measured by sedation (MOAA/S) assessments | up to 480 minutes postdose
Relationships between PK and PD of fospropofol and propofol will be explored using PK/PD modeling. | up to 480 minutes postdose

CONTACTS AND LOCATIONS:
Overall Officials: Talmage Egan, Study Director — Eisai Inc.
Locations (1):
- University of Utah, Salt Lake City Utah, Utah, United States